CLINICAL TRIAL: NCT01375712
Title: Evaluation of the Impact of a Fermented Milk Containing Lactobacillus Casei Strain Shirota on Stool Consistency, Stool Frequency, Constipation-related Symptoms and Quality of Life in People Who Frequently Have Hard or Lumpy Stools
Brief Title: Efficacy Evaluation of Probiotic Product on Bowel Habits in Healthy Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yakult Honsha Co., LTD (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: YAK_BSFS
Record Dates: First submitted 2011-06-15; First posted 2011-06-17 (Estimated); Last update posted 2012-01-31 (Estimated); Status verified 2012-01

CONDITIONS: Constipation
Keywords: Hard or lumpy stools; Stool consistency; Stool frequency; Constipation related symptoms; Constipation related quality of life
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fermented milk (Active Comparator): Fermented milk containing Lactobacillus casei strain Shirota, 65 ml in a bottle, consume 1 bottle per day.
  Interventions: Dietary Supplement: Fermented milk containing Lactobacillus casei strain Shirota
- Placebo (Placebo Comparator): Non-fermented milk without Lactobacillus casei strain Shirota, 65 ml in a bottle, consume 1 bottle per day.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Fermented milk containing Lactobacillus casei strain Shirota — A fermented milk containing Lactobacillus casei strain Shirota, 65 ml for oral administration, 1 bottle per day for 8 weeks (56 days). One bottle of the drink contains: 42.9 kcal/182 kJ; less than 0.1 g of fat; 9.6 g of carbohydrate; 0.01 g of sodium; 0.9 g of protein; and at least 6.5 x 10^9 colony-forming units of Lactobacillus casei strain Shirota.
  Other Names: Commercial name: Yakult
  Arms: Fermented milk
Dietary Supplement: Placebo — Non-fermented milk without Lactobacillus casei strain Shirota, 65 ml for oral administration, 1 bottle per day for 8 weeks (56 days). One bottle of the drink contains: 42.9 kcal/182 kJ; less than 0.1 g of fat; 9.6 g of carbohydrate; 0.01 g of sodium; and 0.9 g of protein.
  Arms: Placebo

SUMMARY:
The objective of this study is to evaluate if consumption of fermented milk containing Lactobacillus casei strain Shirota has an impact on stool consistency, stool frequency, constipation-related symptoms, and quality of life in subjects who frequently have hard or lumpy stools.

DETAILED DESCRIPTION:
Constipation is a common problem affecting approximately 17% of the general population in Europe. Several reports suggest that production of hard or lumpy stools (HLS) is strongly associated with the development of constipation. HLS are produced not only by chronic constipated patient but also by healthy population. Thus, reducing the incidence of HLS might be beneficial in terms of reducing the incidence of constipation in healthy population.

The results of two clinical studies conducted in Europe indicate the positive effect of fermented milk (FM) containing Lactobacillus casei strain Shirota (LcS) to modulate the hardness or dryness of stools. Koebnick et al. (2003) reported that consumption of the FM drink containing LcS decreased the occurrence of hard or lumpy stools, and improved the severity of constipation in patients with chronic constipation in Germany. An open trial conducted in Ghent, Belgium used commercially available FM containing LcS (Yakult® Light) in subjects who frequently had hard or lumpy stools, screened by an average Bristol Stool Form Scale (BS) score < 3.0. After 3 weeks of treatment, the proportion of subjects who produced hard or lumpy stools (BS score = 1 or 2) ≥ 25% of bowel movements decreased from 73.7% at baseline to 36.8%, while in the non-intervention control group the proportion increased from 75.0% to 85.0% during the same period. Based on the results of those studies, it was anticipated that LcS might assist in reducing the production of hard or lumpy stools in the general population. In order to confirm the efficacy in healthy population, a randomised, double blind, placebo control study is required.

ELIGIBILITY:
Inclusion Criteria; a subject:

* is informed both verbally and in writing about the objectives of the clinical study, the methods, the anticipated benefits and potential risks and the discomfort to which he/she may be exposed, and give written consent to participate in the study prior to the start of any study-related procedures
* is healthy female or male, 18-65 years of age, inclusive
* is conscious of having hard or lumpy stools in daily life
* has an average Bristol Stool Form Scale score <3.0 per bowel movement
* female subjects of childbearing potential should use a reliable method of contraception

Exclusion Criteria; a subject:

* is under the age of legal consent
* is mentally or legally incapacitated
* is treated by a doctor for her/his constipation
* has a history of gastrointestinal surgery except for appendectomy
* has a history of chronic gastrointestinal diseases, including but not limited to inflammatory bowel diseases
* has a severe gastrointestinal disorder
* has clinically relevant medical conditions, e.g., renal, hepatic, pulmonary, cardiac, hematological, endocrinological, neurological, or psychiatric conditions
* is pregnant or wanting to become pregnant during the course of the study
* is unable to refrain from or anticipates the use of any medication (including laxatives, diuretics, prescription and non-prescription drugs, vitamins and herbal supplements), except for paracetamol, oral contraceptives, or hormonal replacement therapy during the screening visit and for the duration of the study
* has a history of drug and/or alcohol abuse
* has milk allergies
* is intolerant to lactose

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 238 (Actual)
Dates: Start 2011-06; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Change in the proportion of subjects who produce hard or lumpy stools not less than 25%(≥25%) of weekly number of bowel movements | During pre-treatment (2 weeks) and treatment (8 weeks)
  Hard or lumpy stools are defined as stools with Bristol Stool Form Scale score 1 or 2. Incidence of hard or lumpy stools is calculated by weekly basis.

SECONDARY OUTCOMES:
Weekly average Bristol Stool Form Scale score | During pre-treatment (2 weeks) and treatment (8 weeks)
  Bristol Stool Form Scale is a medical aid designed to classify the form of stool with 7 levels; Separate hard lumps like nuts (difficult to pass), score=1; Sausage-shaped but lumpy, score=2;Like a sausage but with cracks on its surface, score=3; Like a sausage or snake, smooth and soft, score=4; Soft blobs with clear-cut edges (passed easily), score=5; Fluffy pieces with ragged edges, a mushy stool, score=6; Watery, no solid pieces, entirely liquid, score=7.
Weekly number of spontaneous bowel movements | During pre-treatment (2 weeks) and treatment (8 weeks)
  Spontaneous bowel movement is defined as the bowel movements without laxative use
Weekly number of spontaneous complete bowel movements | During pre-treatment (2 weeks) and treatment (8 weeks)
  Spontaneous complete bowel movement is defined as spontaneous bowel movement relieving the feeling of the presence of stool in the distal bowel.
Patient Assessment of Constipation Symptoms (PAC-SYM) score | 6 points (Days 1, 15, 29, 43, 57 and 71)
  PAC-SYM contains 12 questions which are classified into 3 subdomains (stool symptoms, abdominal symptoms, and rectal symptoms). The average scores of total questionnaires and each subdomain are assessed.
Patient Assessment of Constipation Quality of Life (PAC-QOL) score | 6 points (Days 1, 15, 29, 43, 57 and 71)
  PAC-QOL contains 28 questions which are classified into 4 subdomains (physical discomfort, worries and concerns, psychosocial discomfort, and satisfaction). The average scores of total questionnaires and each subdomain are assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Heiko Ilchmann, Principal Investigator — Harrison Clinical Research Deutschland GmbH (Clinical Unit)
Locations (1):
- Harrison Clinical Research Deutschland GmbH, Munich, Germany